CLINICAL TRIAL: NCT05268705
Title: The Impact of Macronutrient Composition on Glucose Dynamics in Everyday Life and During Fasted Cycling in Persons With Type 1 Diabetes
Brief Title: The Impact of Macronutrient Composition on Glucose Dynamics in Persons With Type 1 Diabetes
Acronym: HiLo21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-21042230
Record Dates: First submitted 2022-01-31; First posted 2022-03-07 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: type1diabetes
Keywords: Type 1 diabetes; Nutrition; Exercise; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-carbohydrate-low-fat-low-protein diet (Active Comparator)
  Interventions: Other: 7-day diet
- Low-carbohydrate-high-fat-low-protein diet (Active Comparator)
  Interventions: Other: 7-day diet
- Low-carbohydrate-low-fat-high-protein diet (Active Comparator)
  Interventions: Other: 7-day diet

INTERVENTIONS:
Other: 7-day diet — The participants must follow a 7-day high-carbohydrate-low-fat-low-protein diet before the inclinic study visit at day 8. The in-clinic study visits are identical for all the three study arms.
  Arms: High-carbohydrate-low-fat-low-protein diet
Other: 7-day diet — The participants must follow a low-carbohydrate-high-fat-low-protein diet before the inclinic study visit at day 8. The in-clinic study visits are identical for all the three study arms.
  Arms: Low-carbohydrate-high-fat-low-protein diet
Other: 7-day diet — The participants must follow a low-carbohydrate-low-fat-high-protein diet before the inclinic study visit at day 8. The in-clinic study visits are identical for all the three study arms.
  Arms: Low-carbohydrate-low-fat-high-protein diet

SUMMARY:
A randomized, open-label, three-arm crossover study will be conducted. The aim of the study is to determine the effect of different isocaloric diet macronutrient compositions (High-carbohydrate-Low-fat-Low-protein (HCLFLP), Low-carbohydrate-High-fat-Low-protein (LCHFLP), Low-carbohydrate-Low-fat-High-protein (LCLFHP)) on plasma glucose dynamics in everyday life and during fasted exercise in persons with type 1 diabetes. Our hypothesis is that a HCLFLP diet reduce the decrease in plasma glucose from start to end of fasted exercise compared with a LCHFLP diet. Secondary a LCHFLP compared with a LCLFHP diet does not reduces the decrease in plasma glucose from start to end of fasted exercise. The current study will contribute with new knowledge about the importance of the compositions of a low-carbohydrate diet on glucose dynamics and the influence on plasma glucose during and after cycling in fasted state.

DETAILED DESCRIPTION:
Background:

In order to increase time, spend in euglycemia ranges many persons with type 1 diabetes choose to follow a low-carbohydrate diet. However, to date strong evidence on the effects of low-carbohydrate diets in persons with type 1 diabetes is lacking with even less evidence pertaining around physical activity. Our impression is that many persons with type 1 diabetes follow a low-carbohydrate diet on their own initiative despite published available evidence is sparse. This emphasizes the need for more clinical trials that investigates the glycemic impact of low-carbohydrate diets.

The current guidelines for glucose management during exercise focus on carbohydrate intake and reduction of bolus and/or basal insulin immediately before, during and after exercise. The guidelines only briefly describe low-carbohydrate diet and do not describe matters concerning exercise in fasted state, because of lack of evidence in the field. Exercise in fasted state may be preferable for persons with type 1 diabetes since it increases lipid oxidation and is associated with better glucose stability than nonfasted exercise. Furthermore exercise in fasted state do not increase the risk of hypo- or hyperglycemia compared with a non-exercise control day.

Dietary carbohydrate intake might affect the hepatic glucose response. We will use glucagon as a tool to evaluate the hepatic glucose response after the three different diets.

The current study will contribute new knowledge about the importance of the compositions of a low-carbohydrate diet on glucose dynamics and the influence on plasma glucose during and after cycling in fasted state. In addition, the study will detail the importance of diet carbohydrate content on hepatic glucose response.

Study design:

A randomized, open-label, three-arm crossover study will be conducted, where the participants will serve as their own controls. The participants will complete one screening visit and three different 7-day diet interventions ending with an in-clinic study visit at day 8. The diets will be isocaloric and based on individual energy needs. The compositions will be a HCLFLP, LCHFLP, and a LCLFHP diet. The diet interventions will be in random order and there will be a washout period of 5-35 days.

Diet interventions:

Within a week before day 1 of the diet interventions, the participants must meet at Steno Diabetes Center Copenhagen to be instructed about the forthcoming diet intervention and undergo a physical extermination including weight-, blood pressure- and heart rate meassurement, blood sample collection (albumin, estimated glomerular filtration rate (eGFR), total cholesterol, VLDL, LDL HDL and triglycerides) and a urine sample collection (u-albumin-creatinine-ratio).

The participants must attach and start to use a CGM system the day before the start of the diet interventions (day 0) and a ActiGraph activity sensor in the morning of day 1 of diet interventions. The participants must wear the CGM and activity sensor until the end of the study visit at day 8.

Study visits:

At day 8 the participants must meet in the morning after an overnight fast at Steno Diabetes Center Copenhagen for the study visits. Except for the difference in content of the diets prior to the study visits, the study visits are identical.

After resting for 90 minutes (Observation phase 1), the participants must perform 45 min of cycling on an ergometer bike equaling to 60 % of their peak oxygen consumption or until hypoglycemia (plasma glucose < 3.9 mmol/l) or unbearable symptoms of hypoglycemia (Cycling phase). After cycling the participants are observed for 90 minutes or until hypoglycemia (< 3.9 mmol/l) or unbearable symptoms of hypoglycemia while resting (Observation phase 2). If plasma glucose drops < 3.9 mmol/l or if unbearable symptoms of hypoglycemia occurs during cycling, observation phase 2 or if hypoglycemia (< 3.9 mmol/l) or unbearable symptoms of hypoglycemia has not occurred after 90 min of observation phase 2 150 μg glucagon is given subcutaneously. From injection of glucagon the observation 3 phase begins. The participants will be observed 120 minutes after injection of glucagon. A mixed meal will be served before the participants leave the research facility.

Thoughout the study visits the participants must use their insulin pump. The basalrate will be adjusted according to international guidelines. Blood samples for analyses of glucose, lactate, insulin, glucagon, GLP-1, GIP, ketones, inflammatory markers, cortisol, free fatty acids, growth hormone, albumin, estimated glomerular filtration rate (eGFR), total cholesterol, VLDL, LDL HDL and triglycerides will be drawn. Indirect calorimetry will be performed before, during and after exercise and after injection of glucagon to meassure energy expenditure, respiratory exchange ratio and carbohydrate and lipid oxidation rates. The Borg scale will be used to assess percieved exertion during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type 1 diabetes ≥ 5 years
* Insulin pump use ≥ 1 year
* Use of intermittently scanned continuous glucose monitoring (isCGM) or continuous glucose monitoring (CGM) ≥ 3 months
* HbA1c ≤ 69 mmol/mol (8.5%)
* Self-reported hypoglycemia awareness
* Exercising at least 30 minutes at moderate or vigorous intensity two times per week.

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Use of a hybrid closed-loop system
* Females who are pregnant, breast-feeding or intend to become pregnant during the study period
* Ischemic heart disease
* Severe asthma
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the individual unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the difference between study arms in difference from start to end plasma glucose concentration during 45 min fasted cycling (assessed by YSI (Yellow Spring Instruments 2900 STAT Plus)). | 45 min

SECONDARY OUTCOMES:
Mean CGM glucose level assessed by CGM during diet interventions | 7 days
Time spent < 3.9 mmol/l assessed by CGM during diet interventions | 7 days
Time spent < 3.0 mmol/l assessed by CGM during diet interventions | 7 days
Time spent 3.9-10.0 mmol/l assessed by CGM during diet interventions | 7 days
Time spent > 10.0 mmol/l assessed by CGM during diet interventions | 7 days
Time spent > 13.9 mmol/l assessed by CGM during diet interventions | 7 days
Plasma glucose coefficient of variation assessed by CGM during diet interventions | 7 days
Standard deviation assessed by CGM during diet interventions | 7 days
Number of hypoglycemia events (< 3.9 mmol/l) of at least 15 minutes duration assessed by CGM during diet interventions | 7 days
Energy expenditure after each diet intervention assessed by indirect calorimetry | 15 min
Respiratory exchange ratio after each diet intervention assessed by indirect calorimetry | 15 min
Carbohydrate oxidation rate after each diet intervention assessed by indirect calorimetry | 15 min
Fat oxidation rate after each diet intervention assessed by indirect calorimetry | 15 min
Mean plasma glucose assessed by YSI during cycling and observation phase 2 | 135 min
Plasma glucose nadir assessed by YSI during cycling and observation phase 2 | 135 min
Plasma glucose variation assessed by YSI during cycling and observation phase 2 | 135 min
Plasma glucose standard deviation assessed by YSI during cycling and observation phase 2 | 135 min
Number of hypoglycemia events (< 3.9 mmol/l) assessed by YSI during cycling and observation phase 2 | 135 min
Mean insulin during cycling and observation phase 2 | 135 min
Peak insulin during cycling and observation phase 2 | 135 min
Areal under the curve for insulin during cycling and observation phase 2 | 135 min
Energy expenditure assessed by indirect calorimetry during cycling and observation phase 2 | 135 min
Respiratory exchange ratio assessed by indirect calorimetry during cycling and observation phase 2 | 135 min
Carbohydrate oxidation rate assessed by indirect calorimetry during cycling and observation phase 2 | 135 min
Fat oxidation rate assessed by indirect calorimetry during cycling and observation phase 2 | 135 min
Plasma glucose peak assessed by YSI during observation phase 3 | 120 min
Time to plasma glucose peak assessed by YSI during observation phase 3 | 120 min
Time from glucagon administration to 1.1 mmol/l increase in plasma glucose assessed by YSI during observation phase 3 | 120 min
Change in plasma glucose from injection of glucagon to peak plasma glucose assessed by YSI during observation phase 3 | 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, Professor, Principal Investigator — Steno Diabetes Center Copenhagen, Clinical Reseach, Diabetes Technology Research
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCarthy OM, Kristensen KB, Christensen MB, Schmidt S, Ranjan AG, Nicholas C, Bain SC, Norgaard K, Bracken R. Metabolic and physiological responses to graded exercise testing in individuals with type 1 diabetes using insulin pump therapy. Diabetes Obes Metab. 2023 Mar;25(3):878-888. doi: 10.1111/dom.14938. Epub 2023 Jan 3. PMID 36482870